CLINICAL TRIAL: NCT07115784
Title: Clinical Efficacy of Chlorohexidine Varnish in Reducing Gingival Hyperplasia, Plaque Accumulation, and White-Spot Lesions in Orthodontic Patients: A Split-Mouth Randomised Controlled Trial
Brief Title: Clinical Efficacy of Chlorhexidine Varnish in Reducing Gingival Hyperplasia, Plaque Accumulation, and White Spot Lesions in Orthodontic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Gandhara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/004
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Gingival Hyperplasia; Dental Plaque; Tooth Demineralization
Keywords: Gingival Hyperplasia; Dental Plaque; Enamel decalcification; Gingival overgrowth
MeSH Terms: conditions — Gingival Hyperplasia; Dental Plaque; Tooth Demineralization; Gingival Overgrowth

STUDY DESIGN:
Intervention Model Description: This is a specific type of cross-over design where different interventions are applied to different parts of the mouth in the same individual. Each patient will receive chlorhexidine varnish on one quadrant of the upper arch (experimental group) and placebo on the other quadrant (control group), using random allocation by coin flip.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to the side of varnish application (placebo vs chlorhexidine). Outcomes assessors evaluate standardized photographs and index scores without knowledge of group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine Varnish (Experimental): Participants receive 40% chlorhexidine varnish applied to one upper quadrant. The varnish formulation includes 40% chlorhexidine, 36% sandarac, and 24% ethanol. It is applied using a blunt syringe to the buccal surfaces around orthodontic brackets before bonding and during each monthly follow-up for 3 months. Teeth are dried with compressed air prior to application, and patients are advised not to eat/drink for 3 hours and to avoid brushing until the next day.
  Interventions: Drug: Chlorhexidine Varnish
- Placebo Varnish (Control Arm) (Active Comparator): Participants receive placebo varnish (containing 60% sandarac and 40% ethanol) applied to the opposite upper quadrant using the same technique and schedule as the intervention arm. This serves as the control in the split-mouth design. Patients are blinded to which side received the active or placebo varnish.
  Interventions: Drug: Placebo Varnish

INTERVENTIONS:
Drug: Chlorhexidine Varnish — A 40% chlorhexidine varnish formulation (40% chlorhexidine, 36% sandarac, 24% ethanol) applied topically to the buccal surfaces of teeth in the selected upper quadrant. The varnish is applied using a blunt needle syringe before bonding and at monthly follow-up visits for three months. Teeth are dried before application, and patients are instructed not to eat or drink for 3 hours and to avoid brushing until the next day.
  Arms: Chlorhexidine Varnish
Drug: Placebo Varnish — A placebo varnish composed of 60% sandarac and 40% ethanol applied topically in the same manner and frequency as the chlorhexidine varnish. Used on the opposite quadrant of the same patient in a split-mouth design. Participants are blinded to whether chlorhexidine or placebo was applied.
  Arms: Placebo Varnish (Control Arm)

SUMMARY:
This study investigates whether applying a chlorohexidine varnish (a dental coating) reduces gum overgrowth, plaque buildup, and early tooth decay (white spots) in patients with braces. Each participant's mouth is divided into two sides: one receives the active varnish, and the other receives a placebo. Changes in gum health, plaque, and white spots are tracked over 3 months.

DETAILED DESCRIPTION:
This split-mouth randomized controlled trial evaluates the clinical efficacy of 40% chlorohexidine varnish in reducing gingival hyperplasia, plaque buildup, and white spot lesions (WSLs) among orthodontic patients aged 15-30 years. The study employs a within patient design. Each participant's upper dental arch is divided into contralateral quadrants, randomly assigned (via coin flip) to receive either experimental (40% chlorohexidine varnish) or control (placebo: 60% sandarac/40% ethanol) treatments. The varnish is applied to buccal tooth surfaces and gingival margins at baseline (pre-bonding) and monthly for 3 months. Participants are blinded to treatment assignments and instructed to avoid eating/drinking for 3 hours post-application. Primary outcomes include gingival hyperplasia (Bokenkamp index), plaque accumulation.

The trial targets 22 participants (44 teeth sites), accounting for a 10% non-response rate, recruited from the Orthodontics Department of Sardar Begum Dental College (Peshawar). Exclusion criteria include craniofacial anomalies, pregnancy/lactation, drug allergies ( antibiotics, immunosuppressants), varnish component sensitivity, or mouth breathing. The study addresses a critical need for preventive oral care in orthodontics, where fixed appliances increase plaque retention and demineralization risks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15-30 years
* Subjects of both genders
* Presence of permanent dentition

Exclusion Criteria:

* Craniofacial anomalies (cleft lip or palate)
* Pregnant and lactating mothers
* Patients at higher risk of drug allergies (antibiotics, anticoagulants, immunosuppressants, calcium channel blockers)
* Allergy to any component of the varnishes
* Mouth breathers

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in Gingival Hyperplasia | Baseline (T0) to 3 months (T3)
  Change in gingival hyperplasia score from baseline (T0) to 3 months (T3), assessed using the Bokenkamp index.

SECONDARY OUTCOMES:
Reduction in Plaque Accumulation | Baseline (T0) to 3 months (T3)
  Change in plaque index scores from baseline (T0) to 3 months (T3), using the Silness and Loe Plaque Index.
Reduction in White Spot Lesion Severity | Baseline (T0) to 3 months (T3)
  Change in white spot lesion score from baseline (T0) to 3 months (T3), assessed using the Gorelick Index.

CONTACTS AND LOCATIONS:
Overall Officials: Faryal Haider, Principal Investigator — Sardar Begum Dental College
Locations (1):
- Sardar Begum Dental College & Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including scores for gingival index, plaque index, and white spot lesions, will be made available to qualified researchers upon reasonable request for the purpose of secondary analysis,
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting documents will be available 6 months after publication of the primary results and will remain available for up to 3 years.
Access Criteria: Researchers must submit a written request outlining the purpose of data use, research objectives, and intended outcomes. Requests will be reviewed by the principal investigator and ethics committee. Data will be shared under a data use agreement ensuring confidentiality and ethical use.

REFERENCES:
- [Background] Trombelli L, Farina R, Silva CO, Tatakis DN. Plaque-induced gingivitis: Case definition and diagnostic considerations. J Clin Periodontol. 2018 Jun;45 Suppl 20:S44-S67. doi: 10.1111/jcpe.12939. PMID 29926492
- [Background] Lara-Carrillo E, Montiel-Bastida NM, Sanchez-Perez L, Alanis-Tavira J. Effect of orthodontic treatment on saliva, plaque and the levels of Streptococcus mutans and Lactobacillus. Med Oral Patol Oral Cir Bucal. 2010 Nov 1;15(6):e924-9. doi: 10.4317/medoral.15.e924. PMID 20383105
- [Background] Grover V, Kapoor A, Malhotra R, Battu VS, Bhatia A, Sachdeva S. To assess the effectiveness of a chlorhexidine chip in the treatment of chronic periodontitis: A clinical and radiographic study. J Indian Soc Periodontol. 2011 Apr;15(2):139-46. doi: 10.4103/0972-124X.84383. PMID 21976838
- [Background] Rai P, Pandey RK, Khanna R. Qualitative and Quantitative Effect of a Protective Chlorhexidine Varnish Layer Over Resin-infiltrated Proximal Carious Lesions in Primary Teeth. Pediatr Dent. 2016;38(4):40-5. PMID 27557913
- [Background] Bretz WA, Valente MI, Djahjah C, do Valle EV, Weyant RJ, Nor JE. Chlorhexidine varnishes prevent gingivitis in adolescents. ASDC J Dent Child. 2000 Nov-Dec;67(6):399-402, 374. PMID 11204062
- [Background] Alavi S, Yaraghi N. The effect of fluoride varnish and chlorhexidine gel on white spots and gingival and plaque indices in fixed orthodontic patients: A placebo-controlled study. Dent Res J (Isfahan). 2018 Jul-Aug;15(4):276-282. PMID 30123305